CLINICAL TRIAL: NCT03761056
Title: A Phase 2 Multicenter Study Evaluating the Efficacy and Safety of Axicabtagene Ciloleucel as First-Line Therapy in Subjects With High-Risk Large B-Cell Lymphoma (ZUMA-12)
Brief Title: Study to Evaluate the Efficacy and Safety of Axicabtagene Ciloleucel as First-Line Therapy in Participants With High-Risk Large B-Cell Lymphoma
Acronym: ZUMA-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-112; 2019-002291-13 (EudraCT Number)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — axicabtagene ciloleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleucel (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered.
  Participants who achieve partial response or complete response and subsequently experience disease progression will have an option to receive second course of conditioning chemotherapy therapy and axicabtagene ciloleucel. Participants will receive the same axicabtagene ciloleucel regimen as the original target dose anytime during the study.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: Yescarta®
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
The primary objective of this study is to estimate the efficacy of axicabtagene ciloleucel in participants with high-risk large B-cell lymphoma.

After the end of KTE-C19-112 (ZUMA-12), participants who received an infusion of axicabtagene ciloleucel will complete the remainder of the 15-year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed large B-cell lymphoma
* High-grade large B-cell lymphoma
* Individuals must have a positive interim positron emission tomography (PET) (Deauville PET score of 4 or 5) after 2 cycles (PET2+) of chemoimmunotherapy
* No evidence, suspicion and/or history of central nervous system (CNS) involvement of lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count ≥ 1000/μL
* Platelet count ≥ 75,000/μL
* Absolute lymphocyte count ≥ 100/μL
* Adequate renal, hepatic, pulmonary, and cardiac function defined as:

  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min
  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 upper limit of normal (ULN)
  * Total bilirubin ≤1.5 mg/dL, except in individuals with Gilbert's syndrome
* Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
* No clinically significant pleural effusion
* Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria:

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg cervix, bladder, breast) unless disease free for at least 3 years
* History of Richter's transformation of chronic lymphocytic leukemia or primary mediastinal B-cell lymphoma
* History of autologous or allogeneic stem cell transplant
* Prior CD19-targeted therapy
* Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management
* History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection
* Presence of any indwelling line or drain dedicated central venous access catheters, such as a Port-a-Cath or Hickman catheter, are permitted
* Individuals with detectable cerebrospinal fluid malignant cells, brain metastases, or active CNS lymphoma
* History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
* History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (7):
- United States (5):
  - Banner Health MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Hopital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neelapu SS, Dickinson M, Munoz J, Ulrickson ML, Thieblemont C, Oluwole OO, et al. 739 Primary Analysis of ZUMA-12: A Phase 2 Study of Axicabtagene Ciloleucel (Axi-Cel) As First-Line Therapy in Patients with High-Risk Large B-Cell Lymphoma (LBCL) [Abstract]. 63rd American Society of Hematology (ASH) Annual Meeting and Exposition; 2021 11-14 December.
- [Background] Neelapu SS, Dickinson M, Ulrickson ML, Oluwole OO, Herrera AF, Thieblemont C, et al. 405 Interim Analysis of ZUMA-12: A Phase 2 Study of Axicabtagene Ciloleucel (Axi-Cel) as First-Line Therapy in Patients (Pts) With High-Risk Large B-Cell Lymphoma (LBCL) [Abstract]. 62nd American Society of Hematology (ASH) Annual Meeting and Exposition Virtual; 2020 05-08 December.
- [Background] Neelapu SS, Chavez JC, Lin Y, Munoz J, Ujjani CS, Riedell P, et al. ZUMA-12: A Phase 2 Multicenter Study of Axicabtagene Ciloleucel (Axi-Cel) as a First-Line Therapy in Patients (Pts) with High-Risk Large B-Cell Lymphoma (LBCL) [Abstract]. J Clin Oncol 2019;37 (15).
- [Background] Neelapu SS, Dickinson M, Munoz J, Ulrickson ML, Thieblemont C, Oluwole OO, Herrera AF, Ujjani CS, Lin Y, Riedell PA, Kekre N, de Vos S, Lui C, Milletti F, Dong J, Xu H, Chavez JC. Axicabtagene ciloleucel as first-line therapy in high-risk large B-cell lymphoma: the phase 2 ZUMA-12 trial. Nat Med. 2022 Apr;28(4):735-742. doi: 10.1038/s41591-022-01731-4. Epub 2022 Mar 21. PMID 35314842
- [Background] Chavez JC, Dickinson M, Munoz JL, Ulrickson ML, Thieblemont C, Oluwole OO, et al. 3-Year Analysis of ZUMA-12: A Phase 2 Study of Axicabtagene Ciloleucel (Axi-Cel) As First-Line Therapy in Patients with High-Risk Large B-Cell Lymphoma (LBCL). Blood 2023;142 (Supplement 1):894-7
- [Derived] Chavez JC, Dickinson M, Munoz J, Ulrickson ML, Thieblemont C, Oluwole OO, Herrera AF, Ujjani CS, Lin Y, Riedell PA, Kekre N, de Vos S, Wulff J, Williams CM, Winters J, Kloos I, Xu H, Neelapu SS. Three-year follow-up analysis of first-line axicabtagene ciloleucel for high-risk large B-cell lymphoma: the ZUMA-12 study. Blood. 2025 May 15;145(20):2303-2311. doi: 10.1182/blood.2024027347. PMID 39938019
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, France, and Australia.
Pre-assignment Details: 54 participants were screened.
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered.
  Participants who achieved partial response or complete response and subsequently experienced disease progression had an option to receive second course of conditioning chemotherapy therapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose anytime during the study (Up to 4 years).
Period: Overall Study
Arm/Group | Axicabtagene Ciloleucel
Started | 42
Completed (Completed study and enrolled to long term follow-up (LTFU) protocol, another study (KT-US-982-5968; NCT# NCT05041309).) | 29
Not Completed | 13
Not completed — Death | 8
Not completed — Enrolled but never treated | 2
Not completed — Withdrawal of consent from further follow-up | 2
Not completed — Investigator decision | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered.
  Participants who achieved partial response or complete response and subsequently experienced disease progression had an option to receive second course of conditioning chemotherapy therapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose anytime during the study (Up to 4 years).
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 1
  Race: Black or African American | 1
  Race: White | 33
  Race: Other | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
  France | 2
  Australia | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate Per the Lugano Classification as Determined by Study Investigators
Description: CR Rate is the percentage of participants with CR (complete metabolic response (CMR); complete radiological response (CRR)). CMR: positron emission tomography (PET) 5-point scale (5-PS) scores of 1 (no uptake above background), 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass); no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow (BM). CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion (LDi); no extralymphatic sites of disease; absent non-measured lesion (NMLs); organ enlargement regress to normal; no new sites; and bone marrow normal by morphology.
Time Frame: Up to 4 years
Population: The Response Evaluable Analysis set included participants who were enrolled and treated with axicabtagene ciloleucel at a dose of at least 1 x 10^6 anti-CD19 CAR T cells/kg, and centrally confirmed disease type (double-/triple- hit lymphomas) or International Prognostic Index (IPI) score ≥ 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
percentage of participants | 86 [71 to 95]

2. Secondary Outcome: Objective Response Rate (ORR) Per the Lugano Classification as Determined by Study Investigators
Description: ORR: percentage of participants with CR (CMR;CRR) or PR (partial metabolic response (PMR); partial radiologic response (PRR)). CMR: PET 5PS scores of 1 (no uptake above background, 2 (uptake ≤mediastinum), 3 (uptake >mediastinum but ≤liver) with/without a residual mass; no new lesions; no evidence of FDG-avid disease in BM. CRR: target nodes/nodal masses regressed to ≤1.5 cm in LDi; no extralymphatic sites of disease; absent NMLs; organ enlargement regress to normal; no new sites; bone marrow morphology normal. PMR: scores 4 (uptake moderately >liver),5 (uptake markedly >liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at end of treatment (EOT). PRR: ≥50% decrease in sum of the product of perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites; absent/normal, regressed, but no increase of NMLs; spleen regressed by >50% in length beyond normal; no new sites.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
percentage of participants | 92 [78 to 98]

3. Secondary Outcome: Duration of Response (DOR) Per the Lugano Classification
Description: DOR is defined only for participants who experience an objective response after axicabtagene ciloleucel infusion and is the time from the first objective response to disease progression (PD) (Lugano classification) or death from any cause. Objective response is defined in outcome measure (OM) 2. PD is defined as a score 4 (uptake moderately > liver) or 5 (uptake markedly >liver and/or new lesions) with an increase in intensity of uptake from baseline; new FDG-avid foci consistent with lymphoma at interim or end of treatment assessment; new FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation); new or recurrent FDG-avid foci in bone marrow. Kaplan-Meier (KM) estimates were used for analysis.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set who achieved ORR were analyzed. Participants not meeting the criteria by analysis data cutoff date were censored at their last evaluable disease assessment date prior to the data cutoff date or new anti-lymphoma therapy start (including stem cell transplant or retreatment of axicabtagene ciloleucel), whichever is earlier.
Measure: Median (Full Range); unit: months
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 34
months | NA [NA to NA] — Median, upper and lower limits of confidence interval (CI) were not estimable as participants were censored.

4. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from axicabtagene ciloleucel infusion date to earliest date of disease progression (Lugano classification), commencement of subsequent new anti-lymphoma therapy including stem cell transplant, or death from any cause. PD is defined in OM 3. KM estimates were used for analysis.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set were analyzed. Participants not meeting the criteria by analysis data cutoff date were censored at their last evaluable disease assessment date prior to the data cutoff date.
Measure: Median (Full Range); unit: months
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
months | NA [NA to NA] — Median, upper and lower limits of CI were not estimable as participants were censored.

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from axicabtagene ciloleucel infusion date to the date of disease progression per Lugano classification or death from any cause. PD is defined in OM 3. KM estimates were used for analysis.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set were analyzed. Participants not meeting the criteria by analysis data cutoff date were censored at their last evaluable disease assessment date prior to the data cutoff date or new antilymphoma therapy start date (including stem cell transplant or retreatment of axicabtagene ciloleucel) whichever was earlier.
Measure: Median (Full Range); unit: months
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2 IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered.
  Participants who achieved partial response or complete response and subsequently experienced disease progression had an option to receive second course of conditioning chemotherapy therapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose anytime during the study (Up to 4 years).
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
months | NA [NA to NA] — Median, upper and lower limits of CI were not estimable as participants were censored.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from axicabtagene ciloleucel infusion to the date of death from any cause. KM estimates were used for analysis.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set were analyzed.
Measure: Median (Full Range); unit: months
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered.
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
months | NA [NA to NA] — Median, upper and lower limits of CI were not estimable due to low number of events.

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAE)
Description: An AE was any untoward medical occurrence in a participant in a clinical trial participant, which did not necessarily have a causal relationship with the treatment. Treatment-emergent adverse events were defined as any adverse event with onset on or after the axicabtagene ciloleucel infusion. Serious adverse event was defined as an event that resulted in the following: death; life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital anomaly or birth defect; and medically important event or reaction.
Time Frame: Up to 2 years
Population: Safety Analysis Set included all participants treated with any dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
percentage of participants
  TEAEs | 100
  Treatment-Emergent SAE | 55

8. Secondary Outcome: Percentage of Participants Experiencing Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Value
Description: Grading categories were determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 2 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
percentage of participants
  Hemoglobin | 3
  Alanine Aminotransferase | 8
  Alkaline Aminotransferase | 0
  Aspartate Aminotransferase | 5
  Bilirubin | 20
  Calcium | 5
  Creatinine | 5
  Glucose | 15
  Magnesium | 5
  Sodium | 0
  Urate | 18

9. Secondary Outcome: Percentage of Participants Experiencing Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Decreased Parameter Value
Description: Grading categories were determined by CTCAE version 5.0.
Time Frame: Up to 2 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
percentage of participants
  Hemoglobin | 43
  Leukocytes | 93
  Lymphocytes | 75
  Neutrophils | 95
  Platelets | 25
  Albumin | 3
  Calcium | 10
  Glucose | 0
  Magnesium | 3
  Potassium | 5
  Sodium | 23

10. Secondary Outcome: Relapse With Central Nervous System (CNS) Disease
Description: Relapse with CNS disease was defined as the time from the axicabtagene ciloleucel infusion date to the earliest date of CNS involvement with lymphoma as determined by typical symptoms, cerebrospinal fluid (CSF) evaluation, and/or diagnostic imaging.
Time Frame: Up to 4 years
Population: Participants in the Response Evaluable Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 37
months | 0 [0 to 0]

11. Secondary Outcome: Pharmacokinetics: Peak Level of Anti-CD19 CAR T Cells in Blood
Description: Peak was defined as the maximum number of CAR T cells in blood measured after infusion.
Time Frame: Up to Month 24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
cells/µL | 36.27 [20.51 to 133.96]

12. Secondary Outcome: Peak Serum Level of Granzyme B, Interferon-gamma (IFNg), Interleukin (IL)-2, IL-5, IL-6, IL-8
Description: Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4.
Time Frame: Up to Week 4
Population: Participants in the Safety Analysis Set with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
pg/mL
  Granzyme B | 28.5 [11.8 to 75.6]
  IFNg | 409.4 [157.8 to 856.8]
  IL-2 | 16.4 [9.7 to 32.9]
  IL-5 | 6.3 [6.3 to 26.2]
  IL-6 | 35.1 [13.2 to 181.1]
  IL-8 | 63.0 [30.1 to 107.5]

13. Secondary Outcome: Peak Serum Level of C-Reactive Protein (CRP)
Description: Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4.
Time Frame: Up to Week 4
Population: Participants in the Safety Analysis Set with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
mg/L | 208.4 [60.9 to 407.5]

14. Secondary Outcome: Peak Serum Level of Ferritin
Description: Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4.
Time Frame: Up to Week 4
Population: Participants in the Safety Analysis Set with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
ng/mL | 749.1 [473.9 to 1874.3]

15. Secondary Outcome: Time to Peak Serum Level of Granzyme B, Interferon-gamma (IFNg), Interleukin (IL)-2, IL-5, IL-6, IL-8, CRP, and Ferritin
Description: Time to peak is defined as the number of days from axicabtagene ciloleucel infusion to the date when the cytokine first reached the maximum post-baseline level.
Time Frame: Up to Week 4
Population: Participants in the Safety Analysis Set with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 40
days
  Granzyme B | 8 [8 to 8]
  IFNg | 4 [4 to 8]
  IL-2 | 4 [4 to 4]
  IL-5 | 1 [1 to 4]
  IL-6 | 8 [4 to 8]
  IL-8 | 8 [4 to 8]
  CRP | 4 [4 to 8]
  Ferritin | 8 [6 to 8]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 4 years; Adverse events: Up to 2 years
Description: All-cause mortality: All Enrolled Analysis Set included all enrolled/leukapheresed participants.
  Adverse Events: Axicabtagene Ciloleucel arm: Safety Analysis Set included all participants treated with any dose of study drug.
  Retreatment arm: Safety Retreatment Analysis Set included all participants who underwent retreatment with study drug.
Groups:
- Axicabtagene Ciloleucel: Participants received 500 mg/m^2 cyclophosphamide IV and 30 mg/m^2/day fludarabine IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered.
- Retreatment Axicabtagene Ciloleucel: Participants who achieved partial response or complete response and subsequently experienced disease progression had an option to receive second course of conditioning chemotherapy therapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose anytime during the study (Up to 4 years).
Arm/Group | Axicabtagene Ciloleucel | Retreatment Axicabtagene Ciloleucel
All-Cause Mortality (participants affected / at risk) | 7/42 | 1/1
Serious Adverse Events (participants affected / at risk) | 22/40 | 1/1
Other Adverse Events (participants affected / at risk) | 40/40 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel (N=40) | Retreatment Axicabtagene Ciloleucel (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Covid-19 (Infections and infestations) | 2 | 0
Covid-19 pneumonia (Infections and infestations) | 2 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Periorbital infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 5 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel (N=40) | Retreatment Axicabtagene Ciloleucel (N=1)
Anaemia (Blood and lymphatic system disorders) | 13 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 10 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 20 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 21 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Chills (General disorders) | 11 | 0
Fatigue (General disorders) | 20 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 5 | 0
Pyrexia (General disorders) | 39 | 0
Hypogammaglobulinaemia (Immune system disorders) | 4 | 0
Covid-19 (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 7 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Blood fibrinogen decreased (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 21 | 1
Platelet count decreased (Investigations) | 7 | 0
White blood cell count decreased (Investigations) | 18 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgraphia (Nervous system disorders) | 3 | 0
Encephalopathy (Nervous system disorders) | 8 | 0
Headache (Nervous system disorders) | 28 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 10 | 0
Agitation (Psychiatric disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 11 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 14 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Study Protocol Amendment 2 (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT03761056/Prot_000.pdf
  • Study Protocol: Study Protocol Amendment 3 (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03761056/Prot_003.pdf
  • Statistical Analysis Plan: Statistical analysis plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT03761056/SAP_001.pdf
  • Statistical Analysis Plan: Translational Statistical analysis plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT03761056/SAP_002.pdf